CLINICAL TRIAL: NCT06546878
Title: Cardiac Rehabilitation: Optimisation of the Functional Capacity of Patients Hospitalized With Cardiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José Manuel Afonso Moreira (Other)
Responsible Party: Sponsor-Investigator, José Manuel Afonso Moreira, Clinical Professor, University of Évora
Organization: University of Évora (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Polytechnic Institute of Beja
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Myocardial Ischemia; Heart Diseases
Keywords: Cardiac Rehabilitation; Phase I; Myocardial Ischemia; Rehabilitation Nursing
MeSH Terms: conditions — Myocardial Ischemia; Heart Diseases | interventions — Cardiac Rehabilitation; Clinical Trials, Phase I as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental)
  Interventions: Procedure: Cardiac Rehabilitation (Phase I) - nurse intervention

INTERVENTIONS:
Procedure: Cardiac Rehabilitation (Phase I) - nurse intervention — The intervention consists of applying CR program (phase I ) following the Guidlines of American Association of Cardiovascular and Pulmonary Rehabilitation. The program was applied by adapting it to the patient, varying the intensity and frequency of the sessions, according to the FITT_VP acronym.
  This phase consists of functional respiratory rehabilitation and motor rehabilitation exercises. Each session is divided into three parts, starting with a warm-up with breathing and isometric exercises, then the so-called peak, which consists of specific endurance/aerobic exercises, and at the end, as a recovery phase, relaxation exercises with stretching are instructed.
  Also, health education sessions for patients/caregiver.

SUMMARY:
The World Health Organization [WHO] (2021) states that Cardiovascular Diseases [CVD] are the leading cause of death in the world, and in 2019 around 17.9 million deaths were caused by CVD and the national picture is no different. In Portugal, demographic ageing continues to be established by the increase in average life expectancy, which in turn leads to an increase in the percentage of the population with CVDs. Of particular note is Ischemic Heart Disease [IHD], which is the second leading cause of death in Portugal In order to prevent and combat the progression of CVD and its complications, Cardiac Rehabilitation [CR] programs have emerged as a secondary prevention method supported by relevant scientific evidence. In this sense, the Portuguese Society of Cardiology recognizes the role of the Rehabilitation Nurse Specialist as a crucial element of CR teams.

Objective: To evaluate the effectiveness of the phase I cardiac rehabilitation program in patients hospitalized with ischemic heart disease, in terms of functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Myocardial Ischemia
* Patients who agree to take part in the rehabilitation exercise program
* Patients with the cognitive capacity to understand the instructions given, the exercises to be carried out and the teaching provided
* Patients with clinical and hemodynamic stability
* Patients participating in the rehabilitation exercise program for at least 2 sessions.

Exclusion Criteria:

* Patients who do not meet the safety criteria for exercising after a cardiac event
* Patients with osteoarticular pathology that compromises their ability to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Activity intolerance | The evaluation will be carried out in the first session before starting the rehabilitation program (t0), and in every session during the program for an average of 1 week until the end of the program (t1).
  Modified Borg Dyspnea-It makes it possible to assess the subjective perception of effort and determine safe limits when performing exercises. Esta avaliação permite aos participantes avaliarem-se numa escala de 0 a 10, em que quanto mais baixa for a pontuação, menor será o nível de fadiga.

SECONDARY OUTCOMES:
Health-related quality of life | The evaluation will be carried out in the first session before starting the rehabilitation program (t0). The second evaluation after finishing the program (t1), on average 1 week.
  The EuroQol 5 dimensions (EQ-5D-5L), a two-part instrument, was used to assess HRQoL. It includes a descriptive part with five Likert-type scale questions with response levels (from Level 1 "no problems" to Level 5 "extreme problems") for the five health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The second part reports a visual analog scale (EQ-VAS), scored by the participant by marking an "x" on the scale numbered from 0 ("worst" HRQoL) to 100 ("best" HRQoL), indicating and measuring current general health.
Distance | The first evaluation is carried out in the first session before starting the rehabilitation program (t0), and in all the sessions during the program, on average 1 week before the end of the program (t1).
  Monitoring the distance covered by the patient during the walking phase is fundamental for assessing functional capacity after a cardiac event. The service corridor is wide and 30 meters long and 3 meters wide, marked with tapes on the floor every 3 meters. The distance covered in the service corridor during all the training sessions is recorded in meters.

CONTACTS AND LOCATIONS:
Overall Officials: José Moreira, MsC, Study Chair — University of Évora
Locations (1):
- Beja, Beja, Portugal

IPD SHARING:
Plan to Share IPD: Yes
The selected patients are informed about the program in full and then asked for their questioned about their willingness to participate and recorded on an informed consent form.
  Data collection will be authorized by the participant, following authorization from the Ethics Committee of the Polytechnic Institute of Beja and ULS-Baixo Alentejo.
  They will then be anonymized through coding and stored in a cloud with access only to the SR researcher. The results will then be published in a scientific journal.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be analyzed at the end of the rehabilitation program, and then shared anonymously through publication in a scientific journal.
Access Criteria: Data will only be accessible to researchers associated with the study and will be anonymized, with each participant associated with a coded number.